CLINICAL TRIAL: NCT06801574
Title: EVALUATION OF POSTOPERATIVE EFFECT OF THREE DIFFERENT ANALGESIC TECHNIQUES IN PATIENTS UNDERGOING LUMBAR FIXATION SURGERY USING SALIVARY OPIORPHIN LEVEL: A PROSPECTIVE RANDOMIZED CLINICAL STUDY
Brief Title: Evaluation Of Three Different Anagesic Techniques In Patients Undergoing Lumbar Fixation Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Feyza Şimşek, Dr, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B.30.2.YYU.0.01.00.00/90
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-02

CONDITIONS: Lumbar Fixation Surgery
Keywords: lumbar fixation surgery; erector spinal plane block; local infiltration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Erector Spinae Plane Block (Active Comparator)
  Interventions: Other: Erector Spinae Plane Block
- Group Local Infiltration (Active Comparator)
  Interventions: Other: infiltration
- Group Control (No Intervention)

INTERVENTIONS:
Other: Erector Spinae Plane Block — After the surgical team places the final suture, while the patient is in the prone position, an ultrasound-guided ESP (Erector Spinae Plane) block will be administered bilaterally using a block needle. A total of 40 mL of 0.25% bupivacaine will be injected.
  Arms: Group Erector Spinae Plane Block
Other: infiltration — Before the surgical team closes the incision, local infiltration with 40 mL of 0.25% bupivacaine will be performed at the surgical site.
  Arms: Group Local Infiltration

SUMMARY:
Lumbar spinal stenosis is a degenerative condition characterized by the narrowing of the space surrounding the neurovascular structures of the lumbar vertebrae, resulting from age-related changes in the intervertebral discs, ligamentum flavum, and facet joints. It commonly causes unilateral pain in the lower back, hips, and legs, often described as cramping or burning. Postoperative pain management in these cases frequently involves oral opioids or intravenous administration using patient-controlled analgesia devices. However, opioids are associated with side effects such as reduced gastrointestinal motility, urinary retention, and respiratory depression.

To mitigate these issues, local anesthetic wound infiltration is widely employed by surgeons to manage postoperative pain and reduce opioid consumption following lumbar spinal surgeries.

The primary aim of this study is to compare the postoperative efficacy of three different analgesic methods in patients undergoing elective lumbar fixation surgery, using the percentage change in salivary opiorphin levels as a marker. Additionally, the study seeks to evaluate the correlation between these changes and postoperative pain scores, as well as the amount of opioids consumed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo lumbar fixation surgery under general anesthesia
* aged between 18 and 65 years,
* American Society of Anesthesiologists physical status classification of I-II

Exclusion Criteria:

* Patients with a known allergy to local anesthetics.
* Patients who used opioid analgesics within 48 hours prior to sample collection.
* Patients with a history of smoking or alcohol consumption.
* Patients with conditions affecting salivary flow, such as xerostomia or those who have undergone radiotherapy.
* Patients with infectious diseases known to be transmissible through saliva.
* Patients with an ASA physical status classification of III or higher.
* Patients unable to use a patient-controlled analgesia (PCA) device.
* Patients who do not consent to the study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Postoperative Efficacy of Analgesic Methods Using Salivary Opiorphin Levels | postoperative 24 hours
  The primary aim of this study is to compare the postoperative efficacy of three different analgesic methods applied to patients undergoing elective lumbar fixation surgery by assessing the percentage change in salivary opiorphin levels. Additionally, the study aims to evaluate the correlation of these changes with postoperative Visual Analog Scale (VAS) pain scores and the amount of opioids consumed.

SECONDARY OUTCOMES:
Total amount of opioid consumption | Postoperative 24 hours
  the secondary objective was to measure the total amount of opioid consumption in the first 24 hours postoperatively
Pain scores in first 24 hours at rest and at movement | postoperative 24 hours
  Evaluation of pain scores during movement and rest within 24 hours postoperatively using the Visual Analog Scale
Correlation between basal Salivary Opiorphin Levels and total 24 hours opioid consumption and pain scores | postoperative 24 hours
  The correlation between basal salivary opiorphin levels and total 24-hour opioid consumption, as well as pain scores will be analyzed to reveal any correlation

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Simsek, Principal Investigator — Dr
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Deng K, Huang K, Wu GF. Ultrasound-guided erector spinae plane block in posterior lumbar surgery (Review). Biomed Rep. 2024 Apr 22;20(6):95. doi: 10.3892/br.2024.1783. eCollection 2024 Jun. PMID 38765858
- [Result] Hong B, Baek S, Kang H, Oh C, Jo Y, Lee S, Park S. Regional analgesia techniques for lumbar spine surgery: a frequentist network meta-analysis. Int J Surg. 2023 Jun 1;109(6):1728-1741. doi: 10.1097/JS9.0000000000000270. PMID 36912781
- [Result] Lurie J, Tomkins-Lane C. Management of lumbar spinal stenosis. BMJ. 2016 Jan 4;352:h6234. doi: 10.1136/bmj.h6234. PMID 26727925